CLINICAL TRIAL: NCT01481350
Title: Phase 2 Use of Sildenafil for the Treatment of Post-capillary Hypertension in Patients Undergoing Cardiac Surgery
Brief Title: Sildenafil for Post-capillary Pulmonary Hypertension in Patients Undergoing Cardiac Surgery
Acronym: SiPaHCS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Daniela Pasero, Medical Doctor, University of Turin, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0064280
Record Dates: First submitted 2011-11-25; First posted 2011-11-29 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sildenafil (Experimental): All patient will be treat with a intravenous administration of the drug from the beginning of the intervention, for a maximum of 72 hours.
  Interventions: Drug: sildenafil

INTERVENTIONS:
Drug: sildenafil — The patients will receive a dose of 10 mg every 8 hours, for a maximum time of 72 hours.

SUMMARY:
Pulmonary hypertension increases the perioperative risk in patients undergoing cardiac surgery for valvular heart diseases, especially in patients with a long life mitral valve disease. The present study wants to test the hypothesis that intravenous administration of sildenafil reduces pulmonary vascular resistances and afterload of the right ventricle.

DETAILED DESCRIPTION:
Pulmonary hypertension represents an increased risk for perioperative patients undergoing cardiac surgery for valvular heart disease especially in patients with a long life mitral valve disease complicated by sever pulmonary hypertension, with high risk of developing post operative right ventricular failure during separation from cardiopulmonary by pass. A recent study showed that a single oral administration of sildenafil at the beginning of the cardiac intervention in patients undergoing valvular heart surgery complicated by pulmonary hypertension reduces pulmonary vascular resistances without inducing significant effects on systemic vascular resistances. The present study wants to test the hypothesis that intravenous administration of sildenafil reduces pulmonary vascular resistances and afterload of the right ventricle avoiding right ventricular failure. This should support weaning from cardiopulmonary by pass in patients undergoing cardiac surgery for valvular heart diseases associated to pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing valvular heart surgery associated to post capillary pulmonary hypertension with a mean pulmonary arterial pressure (mPAP)>30mmHg or pulmonary vascular resistance (PVR)>3Wu.

Exclusion Criteria:

* patients younger than 18 years old
* ischemic cardiomyopathy
* Ejection Fraction (EF)<30%
* severe Chronic obstructive pulmonary disease (COPD) with oxygen and bronchodilators therapy
* chronic pulmonary disease, chronic renal failure on dialysis
* hepatic failure
* patients with orotracheal intubation and already admitted to the ICU before the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
reduced mechanical ventilation | seven days
  The primary outcome is the reduction of time on mechanical ventilation

SECONDARY OUTCOMES:
ICU length of stay | 28 days
  The secondary outcome is to evaluate the reduction of intensive care unit length of stay.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Rinaldi, MD, Study Chair — San Giovanni Battista, Hospital University of Turin
Locations (1):
- San Giovanni Battista Hospital University of Turin, Turin, Turin, Italy